CLINICAL TRIAL: NCT03966560
Title: Choroidal Thickness and Its Correlations With Ocular Parameters in Cases With Primary Open-angle Glaucoma
Brief Title: Choroidal Thickness and Its Correlations With Ocular Parameters in Primary Open-angle Glaucoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Afyon Kocatepe University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KAEK-2014/04-74
Record Dates: First submitted 2019-05-16; First posted 2019-05-29 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Glaucoma, Open-Angle
Keywords: choroidal thickness; multifocal electroretinography; optic nerve head; optical coherence tomography; primer open-angle glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Brimonidine Tartrate; dorzolamide; Timolol; Ophthalmic Solutions; brinzolamide; Duotrav; Travoprost; Ganfort; Bimatoprost; Latanoprost

STUDY DESIGN:
Intervention Model Description: prospective controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Primary open-angle glaucoma (Experimental): Participants over 40 years of age and diagnosed with primary open-angle glaucoma.
  Medical treatment was initiated for the diagnosed participants.
  Interventions: Drug: Brimonidine Tartrate; Drug: Dorzolamide (as Dorzolamide Hydrochloride) 20 Mg/mL and Timolol (as Timolol Maleate) 5 Mg/mL Eye Drops; Drug: Brinzolamide/Timolol 10 MG/1 ML-5 MG/1 ML Ophthalmic Suspension; Drug: Travoprost and Timolol; Drug: Bimatoprost and Timolol; Drug: Latanoprost
- Healthy (No Intervention): Healthy volunteers who do not have systemic disease that may affect the choroidal thickness and have no ocular features that may affect test measurements.

INTERVENTIONS:
Drug: Brimonidine Tartrate — Brimonidine tartrate 0.15% 1 eye drop, every day for 6-months
  Other Names: Brimonidine Tartrate 0.15%
  Arms: Primary open-angle glaucoma
Drug: Dorzolamide (as Dorzolamide Hydrochloride) 20 Mg/mL and Timolol (as Timolol Maleate) 5 Mg/mL Eye Drops — Dorzolamide and timolol fixed combination 2 eye drops, every day for 6 months
  Other Names: Dorzolamide and timolol fixed combination
  Arms: Primary open-angle glaucoma
Drug: Brinzolamide/Timolol 10 MG/1 ML-5 MG/1 ML Ophthalmic Suspension — Brinzolamide and timolol fixed combination 2 eye drops, every day for 6 months
  Other Names: Brinzolamide and timolol fixed combination
  Arms: Primary open-angle glaucoma
Drug: Travoprost and Timolol — Travoprost and Timolol fixed combination 1 eye drop, every day for 6 months
  Other Names: Travoprost 0.004%/timolol 0.5% fixed combination
  Arms: Primary open-angle glaucoma
Drug: Bimatoprost and Timolol — Bimatoprost and Timolol fixed combination 1 eye drop, every day for 6 months
  Other Names: Bimatoprost 0.03%/timolol 0.5% fixed combination
  Arms: Primary open-angle glaucoma
Drug: Latanoprost — Latanoprost 0.005% 1 eye drop, every day for 6 months
  Other Names: Latanoprost 0.005%
  Arms: Primary open-angle glaucoma

SUMMARY:
Glaucoma is one of the leading causes of blindness worldwide that is a chronic public health problem. Unfortunately, glaucoma can be diagnosed when the disease reaches a certain level in today's conditions. The aim of this study was to investigate the diagnostic methods that can diagnose glaucoma before it reaches the advanced level and to identify pathophysiological processes. In this study, choroidal thickness was investigated in primary open-angle glaucoma cases and its correlations with OCT and multifocal ERG parameters were evaluated.

DETAILED DESCRIPTION:
In this study, patients with primary open-angle glaucoma who have recently received a new diagnosis with healthy volunteers with age-matched groups were enrolled. All data from 49 glaucoma patients and 47 healthy volunteers were recorded and the study was completed. The study was carried out at the Afyon Kocatepe University Ophthalmology Department between January 2014 and April 2015. Routine ophthalmologic examinations of all participants were performed. Medical treatment was initiated on patients diagnosed with primary open-angle glaucoma. Intraocular pressures and visual acuities of all participants were recorded at baseline, at 1-month, at 3-month, and at 6-month. All participants underwent tests of multifocal electroretinography and the measurements of optic nerve head optical coherence tomography parameters and the choroidal thickness, at the same follow-ups. Visual acuities were measured by using the Snellen chart as the best corrected visual acuity. Intraocular pressures were measured by using applanation tonometry. Choroid thicknesses were also measured and recorded using EDI-OCT mode of optical coherence tomography device (Cirrus HD 4000, Carl Zeiss Meditec AG, Germany). Choroidal thicknesses were measured in three regions: fovea, 3mm nasal and temporal distances of the fovea. The mean of these three measurements was recorded as macular choroidal thickness. The same technician performed all multifocal electroretinography tests of the participants (Metrovision Monpack 3, Metrovision, France). Multifocal electroretinography tests were carried out from a distance of 33 cm using ERG-jet electrode, ground electrode, and a reference electrode. Electrical potential responses from 103 retina regions were recorded. Results were compared statistically and correlations were analyzed (SPSS 20.0, SPSS Inc. IL, USA).

ELIGIBILITY:
Inclusion Criteria for the glaucoma group:

* the best corrected visual acuity (BCVA) of 0.6 and above
* Intraocular pressure being above 21 mmHg
* Detection of open-angle by gonioscopy
* Detection of glaucomatous optic disc pitting by fundus examination
* Visual field defect in perimetry (Carl Zeiss Meditec AG, Germany)

Exclusion Criteria for the glaucoma group:

* A secondary cause of glaucoma
* Angle-closure in gonioscopic examination
* Corneal opacity or cataract at the level that may affect imaging, vitreous pathology
* Intravitreal hemorrhage that may affect fundus appearance, retinal pathology
* Chorioretinopathy, optic neuropathy, optic disc pathology, spherical refractive error of 6D and above, cylindrical refraction error of 3D and above and systemic diseases which may affect ocular blood flow

Inclusion Criteria for the healthy group:

* The best corrected visual acuity (BCVA) of 0.8 and above

Exclusion Criteria for the healthy group:

* Presence of systemic disease that may affect choroid blood flow
* Ocular conditions that may affect test measurements

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Macular choroidal thickness measure | Baseline, 1-month, 3-month, 6-month
  Measuring macular choroidal thickness at baseline, at 1-month, at 3-month and at 6-month by using optical coherence tomography
Changes in multifocal electroretinography parameters (Amplitudes [nv/deg2] and impulse times [ms] of N1, N2 and P1 waves in Ring-1, Ring-2, Ring-3 and Ring-4) | Baseline, 1-month, 3-month, 6-month
  Comparison of the mean multifocal electroretinography parameters (Amplitudes [nv/deg2] and impulse times [ms] of N1, N2 and P1 waves in Ring-1, Ring-2, Ring-3 and Ring-4) at baseline, at 1-month, at 3-month and at 6-month
Changes in amplitudes of N1 wave in Ring-1, Ring-2, Ring-3 and Ring-4 [nv/deg2] | Baseline, 1-month, 3-month, 6-month
  Comparison of the mean amplitudes of N1 wave [nv/deg2] in Ring-1, Ring-2, Ring-3 and Ring-4) at baseline, at 1-month, at 3-month and at 6-month
Changes in amplitudes of N2 wave in Ring-1, Ring-2, Ring-3 and Ring-4 [nv/deg2] | Baseline, 1-month, 3-month, 6-month
  Comparison of the mean amplitudes of N2 wave [nv/deg2] in Ring-1, Ring-2, Ring-3 and Ring-4) at baseline, at 1-month, at 3-month and at 6-month
Changes in amplitudes of P1 wave in Ring-1, Ring-2, Ring-3 and Ring-4 [nv/deg2] | Baseline, 1-month, 3-month, 6-month
  Comparison of the mean amplitudes of P1 wave [nv/deg2] in Ring-1, Ring-2, Ring-3 and Ring-4) at baseline, at 1-month, at 3-month and at 6-month
Changes in impulse times of N1 wave in Ring-1, Ring-2, Ring-3 and Ring-4 [ms] | Baseline, 1-month, 3-month, 6-month
  Comparison of the mean impulse times of N1 wave [ms] in Ring-1, Ring-2, Ring-3 and Ring-4) at baseline, at 1-month, at 3-month and at 6-month
Changes in impulse times of P1 wave in Ring-1, Ring-2, Ring-3 and Ring-4 [ms] | Baseline, 1-month, 3-month, 6-month
  Comparison of the mean impulse times of P1 wave [ms] in Ring-1, Ring-2, Ring-3 and Ring-4) at baseline, at 1-month, at 3-month and at 6-month
Changes in P1/N1 ratio of N2 wave in Ring-1, Ring-2, Ring-3 and Ring-4 | Baseline, 1-month, 3-month, 6-month
  Comparison of the mean P1/N1 ratios of N2 wave in Ring-1, Ring-2, Ring-3 and Ring-4) at baseline, at 1-month, at 3-month and at 6-month
Changes in the mean optic nerve head optical coherence tomography parameters (Retinal nerve fiber layer thickness [micrometers], disc area [mm2], cup-to-disc ratios, cup volume [mm3], neuroretinal rim area [mm2]) | Baseline, 1-month, 3-month, 6-month
  Measuring optic nerve head optical coherence tomography parameters (Retinal nerve fiber layer thickness [micrometers], disc area [mm2], cup-to-disc ratios, cup volume [mm3], neuroretinal rim area [mm2]) at 1-month, at 3-month and at 6-month
Changes in the mean neuroretinal rim area [mm2]) | Baseline, 1-month, 3-month, 6-month
  Measuring neuroretinal rim area [mm2] at 1-month, at 3-month and at 6-month
Changes in the mean cup volume [mm3] | Baseline, 1-month, 3-month, 6-month
  Measuring cup volume [mm3] at 1-month, at 3-month and at 6-month
Changes in the mean cup-to-disc ratios | Baseline, 1-month, 3-month, 6-month
  Measuring cup-to-disc ratios at 1-month, at 3-month and at 6-month
Changes in the mean disc area [mm2] | Baseline, 1-month, 3-month, 6-month
  Measuring disc area [mm2] at 1-month, at 3-month and at 6-month
Changes in the mean retinal nerve fiber layer thickness [micrometers] | Baseline, 1-month, 3-month, 6-month
  Measuring retinal nerve fiber layer thicknesses [micrometers] at 1-month, at 3-month and at 6-month

SECONDARY OUTCOMES:
Best-corrected visual acuity measure | Baseline, 1-month, 3-month, 6-month
  Comparison of the mean best-corrected visual acuities at 1-month, at 3-month and at 6-month
Intraocular pressure measure | Baseline, 1-month, 3-month, 6-month
  Measuring intraocular pressure at 1-month, at 3-month and at 6-month
Correlations between choroidal thickness and other parameters | Baseline, 6-month
  Analyze correlations between changes of choroidal thicknesses and changes of other parameters during the study.